CLINICAL TRIAL: NCT04348838
Title: Prospective Cohort of Patients With Hepatocellular Carcinoma in France
Acronym: CHIEF
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Biobanque de Picardie (Unknown); Société Nationale Française de Gastroentérologie (Other); Association Française pour l'Etude du Foie (AFEF) (Unknown); Federation Francophone de Cancerologie Digestive (Other); Association Nationale des Hépato-Gastroentérologues des Hôpitaux Généraux (ANGH) (Unknown); UNICANCER (Other); Groupe Coopérateur multidisciplinaire en Oncologie (GERCOR) (Unknown); Club de Réflexion des Cabinets et Groupes d'Hépato-Gastroentérologie (CREGG) (Unknown); Association de Chirurgie Hépato-Bilio-Pancréatique et de Transplantation (ACHBT) (Unknown); Société Française de Pathologie (SFP) (Unknown); Société Française de Radiologie (SFR) (Unknown); Societe Francaise de Radiotherapie Oncologique (Other)
Responsible Party: Sponsor
Other Study IDs: PI2019_843_0023
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Cancer of Liver; Hepatocellular Carcinoma
Keywords: cancer; liver; hepatocellular carcinoma; cohort
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Hepatic tissues, blood, urine and stools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatocellular carcinoma (HCC) occurs in 90% of cirrhosis primary liver cancers. In France, 8,500 new cases of HCC occur each year, and about 8,000 deaths per year are related to this cancer. The 5-year survival rate is 10%, one of the lowest survival rates of all cancer types. HCC raises a number of major challenges: HCC is discovered at a curable stage in only 25% of cases, reflecting the marked delay in the diagnosis of early stages. The state of knowledge about HCC is well behind that of other cancers (no biomarker, complex carcinogenesis, influence of the aetiology, poorly valorised data, etc.). Rapid technological progress requires large-scale studies to evaluate new diagnostic and therapeutic modalities.

The CHIEF project constitutes a common basis knowledge for research project using prospectively collected data in patients with HCC, regardless of the cause and stage of the cancer.

This project is a Multicentre longitudinal observational study of patients with HCC with prospective data collection on inclusion and patient follow-up. Constitution of a biological resources collection. 5,000 patients will be included over 2 years with a follow-up of patients of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* New cases of HCC
* suspected case of HCC regardless of the cause, stage, treatment
* Known HCC: drug treatment for recurrence or progression

Exclusion Criteria:

* Associated serious condition threatening life in the short term (with the exception of liver disease itself)
* So-called vulnerable populations: minors, persons under guardianship or temporary guardianship, or person deprived of their liberty by an administrative or judicial decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is including new case patients of HCC regardless of the cause, stage of the disease and treatment, and patients with known HCC.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Variation of progression free survival (PFS) in intent to treat after liver transplantation | from day 1 of inclusion, up to 5 years
  Variation of progression free survival (PFS) in intent to treat after liver transplantation
Variation of time until failure of the strategy after hepatic resection and percutaneous destruction | from day 1 of inclusion, up to 5 years
  Variation of time until failure of the strategy after hepatic resection and percutaneous destruction
Variation of overall survival time (OS) after chemoembolization | from day 1 of inclusion, up to 5 years
  Variation of overall survival time (OS) after chemoembolization
Variation of overall survival time (OS) after radioembolization | from day 1 of inclusion, up to 5 years
  Variation of overall survival time (OS) after radioembolization
Variation of overall survival time (OS) after pharmaceutical treatment | from day 1 of inclusion, up to 5 years
  Variation of overall survival time (OS) after pharmaceutical treatment

SECONDARY OUTCOMES:
Variation of adverse event rate of HCC treatments in clinical practice | from day 1 of inclusion, up to 5 years
  Variation of adverse event rate of HCC treatments in clinical practice
Variation of serious adverse event rate of HCC treatments in clinical practice | from day 1 of inclusion, up to 5 years
  Variation of serious adverse event rate of HCC treatments in clinical practice

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude BARBARE, Pr, Principal Investigator — CHU Amiens; Yves-Edouard HERPE, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No